CLINICAL TRIAL: NCT02090582
Title: Pilot Study on H.O.P.E: Helping Ovarian Cancer Patients Cope During Disease Recurrence
Brief Title: H.O.P.E: Helping Ovarian Cancer Patients Cope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00052239
Record Dates: First submitted 2014-03-04; First posted 2014-03-18 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Platinum-resistant Ovarian Cancer; Recurrent Ovarian Cancer; Palliative Care
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Structured Palliative Care (Other)
  Interventions: Other: Structured Palliative Care
- Usual Care (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Structured Palliative Care — Structured palliative care approach, defined as the gynecologic oncology team performing comprehensive symptom assessment with the Quality Data Collection Tool Palliative Care (QDACT-PC) and providing interventions based on National Comprehensive Cancer Network (NCCN) guidelines. Symptom scores above the acceptable threshold in the QDACT-PC tool that occur after two consecutive visits will automatically trigger palliative care consultation.
  Arms: Structured Palliative Care
Other: Usual Care — Usual care described as current practice by the gynecologic oncology team with referral to PC specialist at provider discretion or at the request of the patient or their families.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to test the effect of the gynecologic oncologists with palliative care specialist collaboration (GO-PC) intervention on patient quality of life.

DETAILED DESCRIPTION:
Eligible patients include women diagnosed with platinum-resistant ovarian cancer or recurrent ovarian cancer cancer. All patient participants will complete two quality of life (QOL) questionnaires and a cost-diary documenting their health care experience at time of consent and every 12 weeks thereafter. Consenting care givers will also be asked to complete two questionnaires to asses the impact of structured palliative care on them every 12 weeks.

Patients will be assigned to two arms randomly: 1) usual care or 2) structured palliative care. The primary endpoint is quality of life. A two-sided Chi-square test will be used to compare the proportion of patients who have improved quality of life after treatment between control arm and intervention arm. The average value of multiple scores after treatment will be used to compare with the baseline score before treatment for each question in the standard questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Platinum-resistant ovarian cancer or recurrent ovarian cancer
* Ability to read and respond to questions in English

Exclusion Criteria:

* Platinum-sensitive recurrent ovarian cancer without a significant clinical event
* Existence of co-morbid disease, which in the opinion of the investigator prohibits participation in the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Quality of Life (Functional Assessment of Cancer Therapy for Ovarian Cancer and Functional Assessment of Chronic Illness Therapy for Palliative Care) | Every 12 weeks for a maximum of 5 years
  A combined FACT-O and FACIT-PAL (version 4)16 will be administered at baseline and 12 week intervals on all subjects. The FACT Measurement System is a validated group of questions that measure health-related QOL in cancer patients. Both questionnaires have identical questions for physical well-being, functional well-being, emotional well-being, and social well-being. The additional subscales of the FACT-O and FACIT-PAL will be combined to provide a comprehensive quality of life assessment specific to ovarian cancer and palliative care.

CONTACTS AND LOCATIONS:
Overall Officials: Paula S Lee, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina